CLINICAL TRIAL: NCT00811837
Title: The Effect of Remifentanil on Established Sunburn-induced Hyperalgesia in Human Volunteers
Acronym: RemiSun 1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Professor Burkhard Gustorff, Medical University of Vienna, Dept. Anaesthesia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RemiSun 1; LS07-040
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Hyperalgesia
Keywords: Sunburn; Remifentanil; Hyperalgesia
MeSH Terms: conditions — Hyperalgesia; Sunburn | interventions — Midazolam; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentail (Experimental): Remifentanil Infusion
  Interventions: Drug: Remifentanil
- Midazolam (Active Comparator): Active Placebo
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Intravenous infusion
  Other Names: Dormicum
  Arms: Midazolam
Drug: Remifentanil — Intravenous infusion
  Other Names: Ultiva
  Arms: Remifentail

SUMMARY:
Treatment of chronic pain is a major clinical challenge since chronic pain is frequent and leads to deterioration of quality of life. An injury or wound can lead to long term changes in the nervous system that make the skin more sensitive at and near the injury; this is termed hyperalgesia and occurs through long term depotentiation (LTP), i.e., a change in the synaptic interaction between neurons.

Opioids are the gold standard for the symptomatic therapy of moderate to severe pain. Now, in animal studies the investigators have discovered previously unrecognized effects of opioids.

UV-B irradaition of the skin of the thigh is an established model of priamary and secondary hyperalgeisa in humans. The investigators want to test the influence of remifentanil, an ultra-short acting opioid, on hyperalgesia observed after UV-B irradiation in human volunteers in a double blind cross-over prospective active placebo controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination
* Drug free for 1 week prior to the study day

Exclusion Criteria:

* Regular use of medication especially analgesics
* Abuse of alcoholic beverages, drug abuse
* History of asthma
* Participation in a clinical trial in the 2 weeks preceding the study
* Symptoms of a clinically relevant illness in the 2 weeks before the first study day
* Resting systolic blood pressure > 135 mmHg or diastolic blood pressure > 85 mmHg
* Acute skin diseases like sunburn on the relevant areas or skin lesions
* Pregnancy or breast feeding
* UV sensitive skin conditions, like Xeroderma pigmentosa

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-07 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Area of pin prick hyperalgesia | 0-6 hours

SECONDARY OUTCOMES:
Stimulus-response (SR) function to a set of modified rigid von Frey filaments (8-512 mN) | 0-6 hours
Heat pain threshold within the area of mechanical hyperalgesia | 0-6 hours
Mechanical pain threshold within the area of pin prick hyperalgesia, area of dynamic allodynia to brush | 0-6 hours
Adverse effects | 30 and 59 min after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Gustorff, MD, Study Chair — Medical University of Vienna
Locations (1):
- Department of Anaesthesia, Medical University of Vienna, Vienna, Austria